CLINICAL TRIAL: NCT02616666
Title: A Pragmatic Randomized Trial to Evaluate the Comparative Effectiveness Between Dapagliflozin and Standard of Care in Type 2 Diabetes Patients (DECIDE Study)
Brief Title: A Pragmatic Randomized Trial to Evaluate the Comparative Effectiveness Between Dapagliflozin and Standard of Care in Type 2 Diabetes Patients
Acronym: DECIDE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: AstraZeneca (Industry); Clinical Practice Research Datalink (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690R00009; 2015-001873-42 (EudraCT Number)
Record Dates: First submitted 2015-11-17; First posted 2015-11-30 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Randomised; Pragmatic; Standard of Care; Dapagliflozin; FORXIGA
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Dapagliflozin 10 mg (Experimental): Patients will be randomized to receive either dapagliflozin or SOC. As this is a pragmatic trial, there will be no additional interventions (apart from collection of PROs and occurrence of hypoglycaemias) and there will be no restriction on how GPs change the randomized treatment regimen (e.g., switch or add drugs). Patients will be followed up for 2 years (+ 12 weeks = 116 weeks) after randomization, regardless of the status of medication.
  Interventions: Drug: Dapagliflozin
- Standard of Care (SOC) (Active Comparator): Patients will be randomized to receive either dapagliflozin or SOC. As this is a pragmatic trial, there will be no additional interventions (apart from collection of PROs and occurrence of hypoglycaemias) and there will be no restriction on how GPs change the randomized treatment regimen (e.g., switch or add drugs). Patients will be followed up for 2 years (+ 12 weeks = 116 weeks) after randomization, regardless of the status of medication.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Dapagliflozin — The product in study is dapagliflozin (FORXIGA™), 10 mg film-coated tablets, and FORXIGA™ should be prescribed according to the instructions in the SmPC and current practice, including up-titration (if considered appropriate by the investigator). Dapagliflozin will be given in combination with metformin.
  Other Names: FORXIGA
  Arms: Dapagliflozin 10 mg
Drug: Standard of Care — The comparator arm consists of SOC. The SOC arm can be sulphonylurea (SU) or non-SU treatments. SU treatments will include any SU and the related insulin secretagogues repaglinide or nateglinide, each of them in combination with metformin. The non-SU treatments can be metformin and dipeptidyl peptidase 4 inhibitors (DPP-4i), or metformin and glitazones (pioglitazone) combination therapy. Other SGLT-2 inhibitors are excluded. All these treatments are approved in the UK for use in this patient population.
  Arms: Standard of Care (SOC)

SUMMARY:
A trial of patients with type 2 diabetes mellitus to evaluate the comparative effectiveness between dapagliflozin and Standard of Care (SOC)

DETAILED DESCRIPTION:
A longitudinal, open labelled, pragmatic randomized 104 week multicentre trial of patients with type 2 diabetes mellitus to evaluate the comparative effectiveness between dapagliflozin and Standard of Care (SOC)

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients should fulfil the following criteria at the time of screening:

1. Provision of informed consent prior to any study specific procedures
2. Females and males aged ≥18 years up to ≤ 75 years
3. Diagnosed with Type 2 Diabetes Mellitus.
4. Uncontrolled on first-line metformin treatment, defined as ≥8 weeks on maximum tolerated dose of metformin and HbA1c > 6.5%.
5. Ability to read and write as judged by the investigator.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment or randomization in the present study
3. Age > 75 years
4. Pregnancy/active breast feeding at the time of inclusion
5. Known moderate to severe renal impairment (eGFR<60ml/min).
6. Participation in an interventional clinical trial ≤ 3 months before enrolment.
7. Unsuitable to participate on mental health grounds, as judged by the investigator.
8. Physician decision to use, as second line treatment, insulin, a GLP1 agonist compound or a SGLT2 inhibitor different from dapagliflozin.
9. Presence of any of the characteristics in which the products in study are contraindicated, as per current labels.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving clinical success as measured by a 4-item composite endpoint. | Assessment of outcome measure will be made at the clinical evaluation that occurs closest to 52 weeks of follow-up (allowing a window of 12 weeks).
  Proportion of patients achieving clinical success as measured by a 4-item composite endpoint including HbA1c reduction vs. baseline (≥ 0.5%), weight loss vs. baseline (≥ 2 Kg), no reported severe or documented hypoglycaemic events since randomization, and no switching from or adding to the treatment to which the patient was randomized (e.g., dapagliflozin or SOC),at the clinical evaluation that occurs closest to 52 weeks of follow-up (allowing a window of 12 weeks).

SECONDARY OUTCOMES:
HbA1c success (HbA1c reduction vs. baseline ≥ 0.5%) at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks). | From randomization to 104 weeks of follow up.
  HbA1c reduction
Weight loss success (weight vs. baseline ≥ 2 Kg) at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks). | closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks)
  Weight Loss success
Severe or documented hypoglycaemic events up to 52 weeks following randomization and separately, up to 104 weeks following randomization (in both cases, allowing a window of 12 weeks). | Up to 52 weeks following randomization and separately, up to 104 weeks following randomization (in both cases, allowing a window of 12 weeks).
  Documented Hypoglycaemic events
To assess differences between dapagliflozin and SOC in the proportion of patients not switching from or adding to the treatment to which the patient was randomized ( | up to 52 weeks following randomization and separately, up to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
  Switching from or adding to the treatment to which the patient was randomized (e.g., dapagliflozin or SOC) up to 52 weeks following randomization and separately, up to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
To assess differences between dapagliflozin and SOC in the change from baseline in HbA1 | HbA1c at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closet to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
  HbA1c at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
To assess differences between dapagliflozin and SOC in the patients worry related to the risk of hypoglycaemic episodes measured b HFS-II Worry Scale at 6,12, 18 and 24 months | At 6, 12, 18 and 24 months
  To assess differences between dapagliflozin and SOC in the patients worry related to the risk of hypoglycaemic episodes measured b HFS-II Worry Scale at 6,12, 18 and 24 months
To assess differences between dapagliflozin and SOC in the patients satisfaction with treatment as measured by the DTSQ at 6, 12, 18 and 24 months | At 6, 12, 18 and 24 months
  To assess differences between dapagliflozin and SOC in the patients satisfaction with treatment as measured by the DTSQ at 6, 12, 18 and 24 months
To assess differences between dapagliflozin and SOC in the patients health related quality of life as measured by SF35v2 at 6, 12, 18 and 24 months | At 6, 12, 18 and 24 months
  To assess differences between dapagliflozin and SOC in the patients health related quality of life, specifically physical, functioning, role functioning and vitality domains as measured by SF35v2 at 6, 12, 18 and 24 months
To assess differences between dapagliflozin and SOC in the proportion of patients needing antihypertensive escalation (dose up titration, switch and add-on strategies), | up to 52 weeks following randomization and separately, up to 104 weeks following randomization.
  Antihypertensive initiation or escalation (dose up titration, switch and add-on strategies), up to 52 weeks following randomization and separately, up to 104 weeks following randomization.
To assess differences between dapagliflozin and SOC in the proportion of patients with diabetic complications: | up to 52 weeks following randomization and separately, up to 104 weeks following randomization.
  Proportion of patients with the following diabetic complications:
  1. Heart failure
  2. Gangrene or amputation of the leg, foot or toe
  3. Diabetic ketoacidosis
  4. Cerebrovascular disease
  5. Nonfatal myocardial infarction
  6. Blindness
  7. Neuropathy
To assess differences between dapagliflozin and SOC in the change from baseline in systolic blood pressure (SBP) (mmHg) and diastolic blood pressure (DBP) (mmHg) | Closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks)
  To assess differences between dapagliflozin and SOC in the change from baseline in systolic blood pressure (SBP) (mmHg) and diastolic blood pressure (DBP) (mmHg) at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
To assess differences between dapagliflozin and SOC in the change from baseline in eGFR | closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
  eGFR (ml/min) at the clinical evaluation that occurs closest to 52 weeks of follow-up and separately, closest to 104 weeks of follow-up (in both cases, allowing a window of 12 weeks).
To assess differences between dapagliflozin and SOC in the healthcare resource utilization up to 52 weeks following randomization and separately, up to 104 weeks following randomization | up to 52 weeks following randomization and separately, up to 104 weeks following randomization.
  Hospitalizations, contacts due to hypoglycaemic events, needing insulin treatment, complications and unscheduled GP visits, up to 52 weeks following randomization and separately, up to 104 weeks following randomization

CONTACTS AND LOCATIONS:
Overall Officials: John Wilding, MBChB, DM, Principal Investigator — Universtiy of Liverpool, University Hospital, Aintree, Longmoor Lane, Liverpool, L9 7AL, UK; Jesús Medina, PhD, Study Director — AstraZeneca; Susan Beatty, MSc, Study Director — Clinical Practice Research Datalink
Locations (132):
- United Kingdom (132):
  - Research Site, Forfar, Angus
  - Research Site, Yate, Avon
  - Research Site, Bracknell, Berkshire
  - Research Site, Reading, Berkshire
  - Research Site, Wokingham, Berkshire
  - Research Site, Alum Rock, Birmingham, Birmingham
  - Research Site, Maesteg, Bridgend
  - Research Site, Chew Stoke, Bristol
  - Research Site, Yate, Bristol
  - Research Site, Iver, Bucks
  - Research Site, Blackwood, Caerphilly
  - Research Site, Hengoed, Caerphilly
  - Research Site, Greenisland, Carrickfergus
  - Research Site, Whitehead, Carrickfergus
  - Research Site, Macclesfield, Cheshire
  - Research Site, Crook, County Durham
  - Research Site, Denbigh, Denbighshire
  - Research Site, Exeter, Devon
  - Research Site, Hull, East Yorkshire
  - Research Site, Romford, Essex
  - Research Site, Pinhoe, Exeter
  - Research Site, Cheltenham, Gloucestershire
  - Research Site, Trafford, Greater Manchester
  - Research Site, Worsley, Greater Manchester
  - Research Site, Alton, Hampshire
  - Research Site, Farnborough, Hampshire
  - Research Site, Gosport, Hampshire
  - Research Site, Havant, Hampshire
  - Research Site, Romsey, Hampshire
  - Research Site, Southampton, Hampshire
  - Research Site, Waterlooville, Hampshire
  - Research Site, Winchester, Hampshire
  - Research Site, Southampton, Hants
  - Research Site, Leominster, Herefordshire
  - Research Site, Fortrose, Highland
  - Research Site, Beckenham, Kent
  - Research Site, Canterbury, Kent
  - Research Site, Faversham, Kent
  - Research Site, Gravesend, Kent
  - Research Site, Rainham, Kent
  - Research Site, Market Square, Kineton, Kineton
  - Research Site, Barnoldswick, Lancashire
  - Research Site, Blackburn, Lancashire
  - Research Site, Darwen, Lancashire
  - Research Site, Lancaster, Lancashire
  - Research Site, Nelson, Lancashire
  - Research Site, Thornton-Cleveleys, Lancashire
  - Research Site, Thornton-Cleveleys, Lancs
  - Research Site, Loughborough, Leicestershire
  - Research Site, Balham, London
  - Research Site, Brockley, London
  - Research Site, London, London
  - Research Site, Rotherhithe, London
  - Research Site, Streatham, London
  - Research Site, Trafford, Manchester
  - Research Site, Liverpool, Merseyside
  - Research Site, Metropolitan Borough of Wirral, Merseyside
  - Research Site, Wembley, Middlesex
  - Research Site, Glyncorrwg, Neath Port Talbot
  - Research Site, Newport, Newport
  - Research Site, Swaffham, Norfolk
  - Research Site, Clevedon, North Somerset
  - Research Site, Pickering, North Yorkshire
  - Research Site, Ripon, North Yorkshire
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Nottingham, Notts
  - Research Site, Bicester, Oxfordshire
  - Research Site, Carterton, Oxfordshire
  - Research Site, Oxford, Oxfordshire
  - Research Site, Wantage, Oxfordshire
  - Research Site, Witney, Oxfordshire
  - Research Site, Oxford, Oxford
  - Research Site, Oxford, Oxon
  - Research Site, Milford Haven, Pembrokeshire
  - Research Site, Tonypandy, Rhondda Cynon Taff
  - Research Site, Pontypridd, Rhondda Cynon Taf
  - Research Site, Telford, Shropshire
  - Research Site, Axbridge, Somerset
  - Research Site, Ayr, South Ayrshire
  - Research Site, Conisbrough, South Yorkshire
  - Research Site, Worsborough, South Yorkshire
  - Research Site, Bury St Edmunds, Suffolk
  - Research Site, Camberley, Surrey
  - Research Site, Guildford, Surrey
  - Research Site, London, Surrey
  - Research Site, Killay, Swansea
  - Research Site, Barry, Vale of Glamorgan
  - Research Site, Nuneaton, Warks
  - Research Site, Alcester, Warwickshire
  - Research Site, Atherstone, Warwickshire
  - Research Site, Bidford-on-Avon, Warwickshire
  - Research Site, Nuneaton, Warwickshire
  - Research Site, Stratford-upon-Avon, Warwickshire
  - Research Site, Warwick, Warwickshire
  - Research Site, Walsall, West Midlands
  - Research Site, Wolverhampton, West Midlands
  - Research Site, Crawley, West Sussex
  - Research Site, Swindon, Wiltshire
  - Research Site, Droitwich, Worcestershire
  - Research Site, Kidderminster, Worcestershire
  - Research Site, Malvern, Worcestershire
  - Research Site, Alton
  - Research Site, Altrincham
  - Research Site, Blackburn
  - Research Site, Cambridge
  - Research Site, Cirencester
  - Research Site, Cockermouth
  - Research Site, Colchester
  - Research Site, Colindale
  - Research Site, Dudley
  - Research Site, Edmonton
  - Research Site, Fareham
  - Research Site, Fleet
  - Research Site, Gravesend
  - Research Site, Hull
  - Research Site, Kings Norton
  - Research Site, Langport
  - Research Site, Liphook
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Maryport
  - Research Site, Morriston
  - Research Site, Oxford
  - Research Site, Petersfield
  - Research Site, Rowlands Castle
  - Research Site, Royal Leamington Spa
  - Research Site, Stansted
  - Research Site, Stratford-upon-Avon
  - Research Site, Torquay
  - Research Site, Wallsend
  - Research Site, Waterlooville
  - Research Site, Wembley